CLINICAL TRIAL: NCT03204123
Title: PSMA PET Imaging of Recurrent Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-306
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Prostate Adenocarcinoma; Prostate Cancer
Keywords: prostate cancer; prostatectomy; biochemical recurrence; Ga-HBED-iPSMA; 16-306
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ga-HBED-iPSMA PET with CT or MRI (Active Comparator): Participants will have a PET scan with Ga-HBED-iPSMA. PET may be combined with CT or MRI at the discretion of the referring clinician.
  Interventions: Drug: Ga-HBED-iPSMA PET; Diagnostic Test: PET/CT; Diagnostic Test: MRI
- Ga-HBED-iPSMA PET with MRI (Active Comparator): Participants will have a PET scan with Ga-HBED-iPSMA and will be combined with MRI. If PET/MR imaging is not available, PET/CT imaging may be substituted. This arm will be closed to accrual and these patients will be analyzed separately.
  Interventions: Drug: Ga-HBED-iPSMA PET; Diagnostic Test: MRI

INTERVENTIONS:
Drug: Ga-HBED-iPSMA PET — Patients will be injected with 100-300 MBq of 68Ga-HBED-iPSMA and after a waiting of 60-90 minutes patients will be scanned from mid-skull to mid-thigh.
Diagnostic Test: PET/CT — PET/CT will be acquired using a GE 710 or 690 time-of-flight PET/CT scanner. Following a waiting period of 60-90 minutes post 68Ga-HBED-iPSMA administration, patients will be scanned from top of the skull to mid-thigh. Images will be acquired with patients in a supine position with their arms raised above their head. If patients cannot raise their arms above the head, the arms will be comfortably positioned and secured by the side of the patient. The PET may be combined with a CT scan as a PET/CT or a MRI scan as PET/MR.
  Arms: Ga-HBED-iPSMA PET with CT or MRI
Diagnostic Test: MRI — Patients may undergo a diagnostic MRI of the prostate, other body parts or a whole-body MRI at the same imaging session as clinically indicated.

SUMMARY:
The purpose of this study is to see if a new diagnostic research agent named 68Ga-HBED-CC-PSMA can show prostate cancer on a PET/CT scan that cannot be seen on other standard imaging even when the PSA levels are very low.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the prostate
* Initially treated with definitive local therapy (surgery and radiation therapy are the most common treatments, but other treatments are also eligible)
* For patients initially treated with surgery, radiation therapy, brachytherapy, or cryotherapy:

  * PSA ≥ 0.2 ng/mL in at least two consecutive tests within 6 months of date of consent for patients
  * Note: The most recent PSA value must be within 6 weeks of consent
* For patients who have received additional treatment in the recurrent or metastatic setting:

  ° PSA ≥ 2 ng/ml above the most recent therapy nadir
* Age ≥ 18 years
* Patient must be able to tolerate PET/CT or PET/MR imaging

Exclusion Criteria:

* Patient with claustrophobia that would preclude PET/CT or PET/MR imaging or other contraindications to CT imaging.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1171 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Disease localization by PSMA PET/MR | 2 years

SECONDARY OUTCOMES:
PSA relapse free survival in patients undergoing PSMA PET/MR guided SRT | 2 years
Incidence of Treatment-Emergent Adverse Events assessed by common terminology criteria for adverse events (CTCAE v4.0) | 2 years
  The safety and tolerability of 68Ga-HBED-iPSMA will be followed by assessing the incidence, nature and severity of toxicities by common terminology criteria for adverse events (CTCAE v4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schöder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/